CLINICAL TRIAL: NCT00277992
Title: Growth in Children With HLHS
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-107
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2007-05-23 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: Pediatric; Cardiac; Norwood operation modification; GT/Nissen operation; Po feed; GT fed
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Children with HLHS have a history of poor enteral intake and growth. Over the past several years a modification to the Norwood operation was instituted (RV to PA shunt in place of the standard Blalock-Taussig shunt).

The purpose of this study is to evaluate whether children who underwent this modification of the Norwood procedure had improved growth compared to those in past years who underwent traditional Norwood.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether children who underwent this modification of the Norwood procedure had improved growth compared to those in past years who underwent traditional Norwood. Also, the standard of care has changed to GT/Nissen operation to facilitate "safe" feeding in those patients who are not able to feed by mouth (po feed).

A second aim of this study is to evaluate whether children who are GT fed have improved growth compared to those who are not.

We wish to review all patients who underwent Norwood procedure from January 1, 2001 to March 31, 2005.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Children's Healthcare of Atlanta, Egleston Norwood procedure between Jan. 1. 2001 and March 31.2005

Exclusion Criteria:

* Those who do not meet inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100
Dates: Start 2001-01

CONTACTS AND LOCATIONS:
Overall Officials: Janet Simsic, MD, Principal Investigator — Children's Healthcare of Atlanta, Sibley Heat Center Cardiology
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States